CLINICAL TRIAL: NCT02654470
Title: Watchman FLX Left Atrial Appendage Closure Device Post Approval Study
Brief Title: Watchman FLX Left Atrial Appendage Closure Device Post Approval Study ( Europe Only)
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Premier Research (Other); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: FLXibility
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Watchman FLX — Patients who are receiving the Watchman FLX device

SUMMARY:
Watchman FLX Left Atrial Appendage Closure Device Post Approval Study

DETAILED DESCRIPTION:
WATCHMAN FLX is intended to prevent thrombus embolization from the left atrial appendage and reduce the risk of life-threatening bleeding events in patients with non-valvular atrial fibrillation who are eligible for anticoagulation therapy or who have a contraindication to anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are eligible for a WATCHMAN FLX device according to current international and local guidelines and currently approved indications;
2. Subject who are willing and capable of providing informed consent and participating in all testing associated with this clinical investigation at an approved clinical investigational centre;
3. Subjects whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the Subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility
2. The subject is unable or not willing to complete follow-up visits and examinations for the duration of the study
3. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion);
4. Documented life expectancy of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who meet all inclusion and no exclusion criteria can be enrolled. A subject who signs informed consent is considered enrolled in the study. The subjects selected for participation will be from the investigator's general patient population.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
procedural success | 7 days post-implant
incidence of stroke, leak, thrombus and death | 1 year
procedural complications | 7-days post implant

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Betts, Principal Investigator — John Radcliffe Hospital, Oxford, UK
Locations (17):
- Aarhus University Hospital, Aarhus, Denmark
- Hospices Civils de Lyon, Lyon, France
- Germany (6):
  - Elisabeth Krankenhaus, Essen
  - Cardio Vasculares Centrum Sankt Katharinen, Frankfurt
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Cardiologicum Hamburg, Hamburg
  - Uni Jena, Jena
  - Herzzentrum Universität Leipzig, Leipzig
- Beaumont Hospital, Dublin, Ireland
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Ospedale San Francesco, Nuoro
- St. Antonius Hospital, Nieuwegein, Netherlands
- Clinical Hospital University of Medicine, Poznan, Poland
- Spain (2):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Virgen Macarena, Seville
- United Kingdom (2):
  - Royal Sussex County Hospital, Brighton
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No